CLINICAL TRIAL: NCT02687451
Title: An Open-Label Single-Dose And Randomized, Double-Blind, Placebo-Controlled Multiple-Dose Study To Evaluate The Efficacy, Safety, Tolerability, And Pharmacokinetics Of Oxymorphone Hydrochloride (HCl) For Acute Moderate To Severe Postoperative Pain In Pediatric Subjects
Brief Title: Clinical Study to Evaluate the Effectiveness, Safety, and Tolerability of Oxymorphone Immediate Release (IR) Oral Liquid in Post Surgical Pediatric Subjects
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Released from PMR
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EN3319-304
Record Dates: First submitted 2016-01-14; First posted 2016-02-22 (Estimated); Results first posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-01

CONDITIONS: Post-Operative Pain; Acute Pain
Keywords: Surgical Pain; Acute Post-Surgical Pain
MeSH Terms: conditions — Pain, Postoperative; Acute Pain | interventions — Oxymorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Oxymorphone HCl Open-Label Phase (Experimental): Oxymorphone HCl Immediate Release Oral Liquid and Oxymorphone HCl Injection; open-label, single-dose, dose selection phase.
  Interventions: Drug: Oxymorphone HCl
- Oxymorphone HCl Multiple-Dose Phase (Experimental): Oxymorphone HCl Immediate Release Oral Liquid and Oxymorphone HCl Injection; placebo controlled, randomized, double-blinded multiple-dose phase.
  Interventions: Drug: Oxymorphone HCl
- Placebo (Placebo Comparator): Sodium Chloride 0.9% solution; comparator for multiple-dose phase.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxymorphone HCl — Oral liquid and injection; dose to be determined by Independent Data Monitoring Committee (IDMC).
  Other Names: Opana
  Arms: Oxymorphone HCl Multiple-Dose Phase; Oxymorphone HCl Open-Label Phase
Drug: Placebo — Placebo Comparator for the double-blinded, placebo-controlled multiple-dose phase.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy, tolerability, safety and pharmacokinetics of Oxymorphone HCl as an analgesic for acute moderate to severe post-operative pain in pediatric subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female <2 years of age at the time of surgery.
2. Must weigh at least 3 kg.
3. Is scheduled to have a surgical procedure for which opioid analgesia will be needed to manage postoperative pain for at least 18 hours following intraoperative and/or postoperative IV analgesia.
4. Is generally healthy as documented by medical history; physical examination (including, but not limited to, the cardiovascular, gastrointestinal, respiratory, and central nervous systems); vital sign assessments; 12-lead electrocardiograms (EKGs); clinical laboratory assessments; and general observations. Any abnormalities or deviations from the acceptable range that might be considered clinically relevant by the study physician or investigator will be evaluated on a case-by-case basis, agreed upon by the Principal Investigator (or sub-investigator), and documented in study files before enrolling the subject in the study.
5. The subject's parent or guardian has been informed of the nature of the study and has provided written informed consent.

   Postoperative:
6. Is anticipated to require an analgesic regimen using a short-acting opioid (non-oxycodone or non-oxymorphone) analgesic after surgery (according to standard of care (SOC) as defined in the protocol).
7. Is an inpatient expected to be hospitalized for 24 hours after dosing with study drug.
8. Has an indwelling access catheter for blood sampling.
9. For Groups A and B: Has demonstrated signs of tolerating oral intake. All infants and children should be able to demonstrate strong suck and swallow reflexes and neurologic alertness and stability sufficient to handle oral secretions.
10. Prior to administration of oxymorphone HCl oral solution, for Groups A and B, had demonstrated the ability to tolerate clear liquids, following surgery according to the SOC at each institution. All infants and children should be able to demonstrate strong suck and swallow reflexes and neurologic alertness and stability sufficient to handle oral secretions. The ability to tolerate small amounts (1 to 2 oz.) of clear liquids without emesis (over 30 to 60 minutes) would support readiness for study participation and oral intake once the physician has ordered the diet advanced to clear liquids and the subject has ingested fluids by mouth without nausea or vomiting.

Exclusion Criteria:

Subjects who meet any of the following criteria will not be eligible to participate in the study:

1. Has the presence or history of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or nervous system(s) or psychiatric disease that would contraindicate participation, as determined by the Investigator.
2. Has any clinical laboratory test result outside the accepted range that has been confirmed upon re-examination and deemed to be clinically significant.
3. Has a clinically significant illness or condition any time before dosing with study drug that would contraindicate participation, as determined by the Investigator.
4. Has a life expectancy <8 weeks.
5. For age groups A and B: Has a malabsorption, gastroenterologic, or abdominal condition that would interfere with the absorption of study drug.
6. Has evidence of increased intracranial pressure.
7. Has a respiratory condition requiring intubation or resulting in active bronchiolitis, asthma, stridor, or difficulty breathing due to congestion and increased nasal secretions, including oxygen (O2) saturation ≤92%.
8. Has a history of seizures.
9. Subject (and/or mother if subject is nursing) has used medications with actions characteristic of monoamine oxidase inhibitors (MAOIs) within 14 days before the start of the study drug is prohibited. Standard daily pediatric multivitamins may be taken until enrollment into the study but will be restricted during the study.
10. Subject (and/or mother if subject is nursing) has received preoperative opioids for more than 72 consecutive hours.
11. Subject (and/or mother if subject is nursing) has received oxycodone or oxymorphone within 48 hours prior to screening.
12. Subject (and/or mother if subject is nursing) has ingested caffeine- or xanthine-containing products (eg, theophylline) within 48 prior to screening. These products are also prohibited during periods when blood samples are collected.
13. Has a history of relevant drug allergies, food allergies, or both (ie, allergy to oxymorphone or other opioid analgesics) that could interfere with the study.
14. Parent or legal guardian is unable to provide consent for any reason (eg, mental or physical disabilities, language barriers, or is unavailable).
15. Subject (and/or mother if subject is nursing) has participated in a clinical study of an unapproved drug within the previous 30 days.
16. Is not suitable for entry into the study in the opinion of the Investigator.

Ages: 0 Years to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Dalton, Study Director — Endo Pharmceuticals
Locations (3):
- United States (3):
  - Endo Clinical Trial Site #2, Durham, North Carolina
  - Endo Clinical Trial Site #1, Dallas, Texas
  - Endo Clinical Trial Site #4, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A (6 Months - <2 Years) 0.05 mg/kg; Group A (6 Months - <2 Years) 0.10 mg/kg; Group A (6 Months - <2 Years) 0.15 mg/kg; Group B (61 Days - <6 Months) 0.10 mg/kg: Oxymorphone HCl Immediate Release Oral Liquid and Oxymorphone HCl Injection; open-label, single-dose, dose selection phase.
- Oxymorphone HCl Multiple Dose Phase (6 Months - <2 Years): Oxymorphone HCl Immediate Release Oral Liquid and Oxymorphone HCl Injection.
- Placebo: Sodium Chloride 0.9%; comparator for multiple dose phase.
Period: Overall Study
Arm/Group | Group A (6 Months - <2 Years) 0.05 mg/kg | Group A (6 Months - <2 Years) 0.10 mg/kg | Group A (6 Months - <2 Years) 0.15 mg/kg | Group B (61 Days - <6 Months) 0.10 mg/kg | Oxymorphone HCl Multiple Dose Phase (6 Months - <2 Years) | Placebo
Started | 6 | 5 | 5 | 5 | 4 | 3
Completed | 5 | 5 | 5 | 5 | 4 | 2
Not Completed | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (6 Months - <2 Years) 0.05 mg/kg | Group A (6 Months - <2 Years) 0.10 mg/kg | Group A (6 Months - <2 Years) 0.15 mg/kg | Group B (61 Days - <6 Months) 0.10 mg/kg | Oxymorphone HCl Multiple Dose Phase (6 Months - <2 Years) | Placebo | Total
Number analyzed (Participants) | 6 | 5 | 5 | 5 | 4 | 3 | 28
Age, Continuous [Mean (Standard Deviation); unit: Days] — Population: Single Dose Safety Population and Multiple Dose Safety Population
  Days
    Single Dose Safety Population: number analyzed (Participants) | 6 | 5 | 5 | 5 | 0 | 0 | 21
    Single Dose Safety Population | 384.2 (106.83) | 295.2 (84.19) | 466.4 (128.76) | 108.4 (11.72) |  |  | 316.9 (159.83)
    Multiple Dose Safety Population: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 3 | 7
    Multiple Dose Safety Population |  |  |  |  | 396.5 (129.88) | 627.0 (75.11) | 495.3 (159.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 3 | 2 | 2 | 1 | 14
  Male | 2 | 3 | 2 | 3 | 2 | 2 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 4 | 2 | 3 | 1 | 11
  Not Hispanic or Latino | 5 | 5 | 1 | 3 | 1 | 2 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 1 | 0 | 0 | 0 | 5
  White | 4 | 3 | 4 | 3 | 4 | 3 | 21
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 0 | 0 | 2
Weight [Mean (Standard Deviation); unit: Kg] — Population: Single Dose Safety Population and Multiple Dose Safety Population
  Kg
    Single Dose Safety Population: number analyzed (Participants) | 6 | 5 | 5 | 5 | 0 | 0 | 21
    Single Dose Safety Population | 9.39 (0.855) | 9.48 (1.442) | 10.14 (1.841) | 5.95 (0.877) |  |  | 8.77 (2.031)
    Multiple Dose Safety Population: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 3 | 7
    Multiple Dose Safety Population |  |  |  |  | 9.33 (1.797) | 11.53 (2.079) | 10.27 (2.109)
Height [Mean (Standard Deviation); unit: cm] — Population: Single Dose Safety Population and Multiple Dose Safety Population
  cm
    Single Dose Safety Population: number analyzed (Participants) | 6 | 5 | 5 | 5 | 0 | 0 | 21
    Single Dose Safety Population | 72.72 (2.129) | 72.28 (3.943) | 74.60 (6.387) | 59.00 (3.921) |  |  | 69.80 (7.382)
    Multiple Dose Safety Population: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 3 | 7
    Multiple Dose Safety Population |  |  |  |  | 74.25 (6.551) | 83.00 (1.732) | 78.00 (6.658)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: Single Dose Safety Population and Multiple Dose Safety Population
  kg/m^2
    Singe Dose Safety Population: number analyzed (Participants) | 6 | 5 | 5 | 5 | 0 | 0 | 21
    Singe Dose Safety Population | 17.73 (1.496) | 18.04 (0.904) | 18.12 (1.156) | 17.10 (1.804) |  |  | 17.75 (1.343)
    Multiple Dose Safety Population: number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 3 | 7
    Multiple Dose Safety Population |  |  |  |  | 16.83 (1.841) | 16.73 (2.775) | 16.79 (2.065)

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Total Amount of Morphine Rescue Medication Required for Analgesia in the Active Treatment Group (Single Dose)
Time Frame: Up to 24 hours post dose
Population: Single Dose Safety Population
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Group A (6 Months - <2 Years) 0.05 mg/kg | Group A (6 Months - <2 Years) 0.10 mg/kg | Group A (6 Months - <2 Years) 0.15 mg/kg | Group B (61 Days - <6 Months) 0.10 mg/kg
Number analyzed (Participants) | 4 | 5 | 1 | 4
mg | 3.348 (3.0745) | 1.886 (1.5034) | 1.400 (NA) — Only one observation; therefore Standard Deviation (SD) cannot be calculated | 0.725 (0.3797)

2. Secondary Outcome: Assessment of Pain Using the Age Appropriate Scale, Face, Legs, Activity, Cry, Consolability (FLACC) or the Neonatal Infant Pain Scale (NIPS).
Description: The Face, Legs, Activity, Cry, Consolability (FLACC) was used for patients between the ages of 6 months and 2 years. The FLACC scale is a validated scale that measures pain in patients who are awake or asleep based on a composite score of observations of facial expression, tonicity in legs, activity scores, the presence of crying, and whether the participant is consolable. Each category is scored on a 0 to 2 scale, which results in a total possible score of 0-10. Assessment of the behavioral score are relaxed and comfortable (0), mild discomfort (1-3), moderate pain (4-6), and severe discomfort/pain (7-10). The Neonatal Infant Pain range from 0-7 The NIPS was used for patients 0 to < 6 months.
Time Frame: Single Dose Phase: at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6 and 8 hours post dose. Multiple Dose Phase: every 0.5 hours up to 24 hours post first dose.
Population: Single Dose Phase: Evaluable population =all subjects who received at least 1 dose of drug and provided at least 4 hrs of post-dose assessments and at least 3 PK assessments. Multiple dose Phase: Intent to-treat (ITT) population =all randomized subjects who received at least 1 dose of study drug and completed at least 1 post-dose pain intensity assessment. Due to safety concerns, raised by the IDMC, efficacy analyses were not conducted.
Arm/Group | Group A (6 Months - <2 Years) 0.05 mg/kg | Group A (6 Months - <2 Years) 0.10 mg/kg | Group A (6 Months - <2 Years) 0.15 mg/kg | Group B (61 Days - <6 Months) 0.10 mg/kg | Oxymorphone HCl Multiple Dose Phase (6 Months - <2 Years) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Pharmacokinetic Variable: Volume of Distribution (Vd)
Time Frame: Single Dose Phase: at 0 (Baseline), 0.5, 1.0, 2.0, 3.0, 4.0, 8.0, and 24 hours post dose. Multiple Dose Phase: Baseline before each dose only
Population: The PK (Pharmacokinetic) population included all patients who received oxymorphone HCl (immediate-release oral liquid or IV formulation) and had plasma concentration data from at least 1 time point from either single-dose or multiple-dose phase to facilitate the population PK modeling and analysis. The study was terminated early due to safety concerns raised by the IDMC, only the planned safety analyses as specified in the statistical analysis plan were conducted.
Arm/Group | Group A (6 Months - <2 Years) 0.05 mg/kg | Group A (6 Months - <2 Years) 0.10 mg/kg | Group A (6 Months - <2 Years) 0.15 mg/kg | Group B (61 Days - <6 Months) 0.10 mg/kg | Oxymorphone HCl Multiple Dose Phase (6 Months - <2 Years) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Pharmacokinetic Variable: Clearance (CL)
Time Frame: Single Dose Phase: at 0 (Baseline), 0.5, 1.0, 2.0, 3.0, 4.0, 8.0, and 24 hours post dose. Multiple Dose Phase: Baseline before each dose
Population: The PK population included all patients who received oxymorphone HCl (immediate-release oral liquid or IV formulation) and had plasma concentration data from at least 1 time point from either single-dose or multiple-dose phase to facilitate the population PK modeling and analysis. The study was terminated early due to safety concerns raised by the IDMC, only the planned safety analyses as specified in the statistical analysis plan were conducted.
Arm/Group | Group A (6 Months - <2 Years) 0.05 mg/kg | Group A (6 Months - <2 Years) 0.10 mg/kg | Group A (6 Months - <2 Years) 0.15 mg/kg | Group B (61 Days - <6 Months) 0.10 mg/kg | Oxymorphone HCl Multiple Dose Phase (6 Months - <2 Years) | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Cumulative Total Amount of Morphine Rescue Medication Required for Analgesia in the Active Treatment Group Versus Placebo Group (Multiple Dose).
Time Frame: Up to 24 hours post dose
Population: Multiple Dose Safety Population
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Oxymorphone HCl Multiple Dose Phase (6 Months - <2 Years) | Placebo
Number analyzed (Participants) | 0 | 1
mg |  | 0.80 (NA) — Only one observation; therefore Standard Deviation (SD) cannot be calculated

ADVERSE EVENTS:
Time Frame: Time of informed consent through 14 days after the last dose
Description: All serious and non-serious AEs, whether elicited or observed during study visit or spontaneously reported by the participant, including events that occurred from the time the participant signed the study specific consent form until completion of or discharge from the study
Arm/Group | Group A (6 Months - <2 Years) 0.05 mg/kg | Group A (6 Months - <2 Years) 0.10 mg/kg | Group A (6 Months - <2 Years) 0.15 mg/kg | Group B (61 Days - <6 Months) 0.10 mg/kg | Oxymorphone HCl Multiple Dose Phase (6 Months - <2 Years) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/5 | 0/5 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 1/5 | 0/5 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 4/6 | 2/5 | 5/5 | 2/5 | 1/4 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (6 Months - <2 Years) 0.05 mg/kg (N=6) | Group A (6 Months - <2 Years) 0.10 mg/kg (N=5) | Group A (6 Months - <2 Years) 0.15 mg/kg (N=5) | Group B (61 Days - <6 Months) 0.10 mg/kg (N=5) | Oxymorphone HCl Multiple Dose Phase (6 Months - <2 Years) (N=4) | Placebo (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (6 Months - <2 Years) 0.05 mg/kg (N=6) | Group A (6 Months - <2 Years) 0.10 mg/kg (N=5) | Group A (6 Months - <2 Years) 0.15 mg/kg (N=5) | Group B (61 Days - <6 Months) 0.10 mg/kg (N=5) | Oxymorphone HCl Multiple Dose Phase (6 Months - <2 Years) (N=4) | Placebo (N=3)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 4 (7) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (3) | 1 (1) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Post procedural oedema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Incision site swelling (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trismus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT02687451/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/51/NCT02687451/SAP_001.pdf